CLINICAL TRIAL: NCT05763849
Title: A Confirmatory Efficacy Study of Interoceptive Exposure for Adolescents With Low Weight Eating Disorders
Brief Title: Interoceptive Exposure for Adolescents With Low Weight Eating Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Tom Hildebrandt, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-22-01323; 1R01MH131655 (NIH)
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Intervention Model Description: This RCT includes a parallel group design including two psychological treatments (Exposure-based Family Therapy vs. Family Based Therapy) for low weight eating disorders with 12 month follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interoceptive Exposure Treatment (IE) (Experimental): Interoceptive Exposure Therapy (IE) targets food avoidance, food exposure, and body image exposure.
  Interventions: Behavioral: Interoceptive Exposure Treatment (IE)
- Family-Based Treatment (FBT) (Active Comparator): Family-Based Therapy (FBT) focuses on parent-enforced contingencies, increasing value of eating, and decreasing the value of food avoidance.
  Interventions: Behavioral: Family-Based Treatment (FBT)

INTERVENTIONS:
Behavioral: Interoceptive Exposure Treatment (IE) — Interoceptive Exposure Therapy (IE) targets food avoidance in Anorexia Nervosa. Each session the therapist weighs the patient, checks-in, and reviews weekly homework. Sessions occur weekly for 20 weeks, with the first session lasting 1.5 hours and the remaining sessions one hour. Early sessions include using exposure to foods and counterconditioning to pair a positive stimulus with a food that would typically produce food avoidance. Parents are trained to model this at home. Sessions mid-way through address the use of non-judgmental description of appearance during mirror exposure. Sessions at the end of the 20 weeks are focused on recognizing change, planning for future obstacles, and developing a relapse prevention plan to continue practicing distress tolerance, counter-conditioning, and food/body exposure.
  Arms: Interoceptive Exposure Treatment (IE)
Behavioral: Family-Based Treatment (FBT) — Family-Based Therapy (FBT) includes parent-enforced contingencies to increase value of eating and decrease the value of food avoidance. Each session the therapist weighs the patient, checks-in, and reviews weekly homework. Sessions occur weekly for 20 weeks, with the first session lasting 1.5 hours and the remaining sessions one hour. Sessions consist of checking in with the patient, discussion of the week's implementation of refeeding, and helping parents separate the illness from their child. In session 2, a family meal provides the therapist with an opportunity for direct observation of the familial interaction patterns around eating. The therapist makes careful and persistent requests for united parental action toward re-feeding and/or regulating eating habits, the primary concern at this point of the treatment, and the therapist tries to create and reinforce a strong parental alliance around efforts at feeding the child.
  Arms: Family-Based Treatment (FBT)

SUMMARY:
This project includes a parallel group randomized controlled trial comparing two psychological treatments: 1) Exposure-based Family Therapy (IE) vs. 2) Family Based Therapy (FBT) for low weight eating disorders with 12 month follow-up. Primary outcomes are expected body weight and clinical impairment. Three mechanisms of change (Autonomous Eating, Non-Judgmental Body Awareness, and Extinction Learning) will be examined in a process mediation models of change.

DETAILED DESCRIPTION:
A total of 120 individuals with Anorexia Nervosa ages 12-18 will be enrolled to either 20 sessions of outpatient Exposure-based Family Therapy (IE) or Family Based Therapy (FBT). The aims of the study are to test the comparative efficacy and primary mechanisms of change after 6 months of treatment and at one year post-treatment and to explore the mediators and moderators of the primary outcomes at these endpoints. All recruitment and study procedures will take place through the Center of Excellence in Eating and Weight Disorders at the Icahn School of Medicine at Mount Sinai. Assessments will take place at 2-, 4-, 6-, 12-, and 18-months following baseline.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12-18
* Speak English
* Permission from pediatrician or equivalent to receive outpatient care
* Clinically significant restriction of food intake by EDA-5 or evidence of persistent food avoidance from patient or guardians
* Evidence of the inability to maintain greater than minimally low body weight based on BMI for age percentiles and growth trajectories

Exclusion Criteria:

* Comorbid psychotic or bipolar disorder
* Active suicidal ideation
* Current substance dependence
* Psychiatric medication initiated or dosage changes <2 weeks from baseline
* Major medical illness (e.g., diabetes mellitus, Crohn's disease, etc.)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in Expected Body Weight Percentage | Baseline and 6-months
  Expected body weight percentage will be calculated at baseline and end of treatment (6-months) to calculate difference.
Change in Expected Body Weight Percentage | Baseline and 18-months
  Expected body weight percentage will be calculated at baseline and 1 year after treatment (18-months) to calculate difference.
Change in Impairment | Baseline and 6-months
  Impairment is measured using the Clinical Impairment Assessment, which is a 16-item self-report measure of impairment from eating disorders. Responses are scored using 0, 1, 2, or 3 and the score is calculated using the sum of all items. Possible scores range between 0 - 48, with higher scores indicating more impairment and lower scores indicating less impairment. Change in impairment will be calculated using the baseline and end of treatment (6-months) scores from CIA.
Change in Impairment | Baseline and 18-months
  Impairment is measured using the Clinical Impairment Assessment, which is a 16-item self-report measure of impairment from eating disorders. Responses are scored using 0, 1, 2, or 3 and the score is calculated using the sum of all items. Possible scores range between 0 - 48, with higher scores indicating more impairment and lower scores indicating less impairment. Change in impairment will be calculated using the baseline and 1 year after treatment (18-months) scores from CIA.

SECONDARY OUTCOMES:
Change in Autonomous Eating | Baseline and 6-months
  Autonomous eating will be measured in total calories consumed during a single-item meal. Change in total calories consumed will be calculated between baseline and end of treatment (6-months).
Change in Autonomous Eating | Baseline and 18-months
  Autonomous eating will be measured in total calories consumed during a single-item meal. Change in total calories consumed will be calculated between baseline and 1 year after treatment (18-months).
Change in Food Cue Learning | Baseline and 6-months
  Food cue learning is a task completed on a computer that tests associations between food and level of disgust. Pictures of food are shown including fresh and rotten versions of each and participants then rate on a scale from yucky to yummy for each. These ratings produce an extinction rate. There is no set range for scoring, however lower rates indicate more impairment and higher rates indicate less impairment. Extinction rate will be calculated between baseline and end of treatment (6-months).
Change in Food Cue Learning | Baseline and 18-months
  Food cue learning is a task completed on a computer that tests associations between food and level of disgust. Pictures of food are shown including fresh and rotten versions of each and participants then rate on a scale from yucky to yummy for each. These ratings produce an extinction rate. There is no set range for scoring, however lower rates indicate more impairment and higher rates indicate less impairment. Extinction rate will be calculated between baseline and 1 year after treatment (18-months).
Change in Eating Disorder Symptoms | Baseline and 6-months
  Youth Eating Disorder Questionnaire (Y-EDE-Q) is a self-report measure assessing psychopathology of eating disorders in youth using 39 items. Global scores range from 0 to 6 with higher scores indicating symptoms of higher severity. Scores will be calculated between baseline and end of treatment (6-months).
Change in Eating Disorder Symptoms | Baseline and 18-months
  Youth Eating Disorder Questionnaire (Y-EDE-Q) is a self-report measure assessing psychopathology of eating disorders in youth using 39 items. Global scores range from 0 to 6 with higher scores indicating symptoms of higher severity. Scores will be calculated between baseline and end of treatment (6-months).
Change in Nonjudgmental Body Awareness | Baseline and 6-months
  Body awareness Questionnaire (BAQ) is a self-report measure assessing awareness of body sensitivity and changes using 18 items on a score range of 18-126. Higher scores indicate more awareness of body regulation. Scores will be calculated between baseline and end of treatment (6-months).
Change in Nonjudgmental Body Awareness | Baseline and 18-months
  Body awareness Questionnaire (BAQ) is a self-report measure assessing awareness of body sensitivity and changes using 18 items on a score range of 18-126. Higher scores indicate more awareness of body regulation. Scores will be calculated between baseline and end of treatment (18-months).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hildebrandt, Psy.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Department of Psychiatry, Eating and Weight Disorders Program, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Specify Other Time FrameTwice yearly and for each publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.
  Any purpose. Specify Other Mechanism Data will be made available through the National Institute of Mental Health Data Archive (NDA)